CLINICAL TRIAL: NCT01717989
Title: Study to Evaluate the Prospective Payment System Impact on Small Dialysis Organizations
Brief Title: Study to Evaluate the Prospective Payment System
Acronym: STEPPS™
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20080234
Record Dates: First submitted 2012-09-12; First posted 2012-10-31 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Kidney Disease
Keywords: Dialysis; Prospective Payment System; Center for Medicare and Medicaide Services; End Stage Renal Disease; Concomitant Medications Dosage /Treatment patterns
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients with end-stage renal disease (ESRD) treated at small dialysis organizations (SDOs).

SUMMARY:
To describe trends in treatment patterns of Small Dialysis Organizations (SDOs) prior to and during the implementation of the Centers for Medicare and Medicaid Services' (CMS') policy [End Stage Renal Disease (ESRD) Prospective Payment System (PPS)] to bundle reimbursement for all dialysis services. Specifically, to describe CMS ESRD PPS quality performance measures for dialysis centers over time.

ELIGIBILITY:
Patient Inclusion Criteria:

* Adults ≥ 18 years of age who have given written informed consent
* Documented physician diagnosis of ESRD requiring dialysis and receiving care at a participating dialysis center
* Undergoing dialysis on the dialysis schedule assigned to the site

Patient Exclusion Criteria:

* Patients will be ineligible for the study if they do not consent to have their data collected for research purposes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 50 SDOs selected to participate in the registry. All efforts will be made to select a diversified group of facilities by evaluating geography, facility size (i.e., number of patients treated) and setting (i.e., rural and urban settings) and potentially, dialysis modalities offered as well as payor mix.
Sampling Method: Non-Probability Sample
Enrollment: 2248 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (36):
- United States (35):
  - Research Site, Gulf Shores, Alabama
  - Research Site, Siloam Springs, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Covina, California
  - Research Site, Glendale, California
  - Research Site, Hacienda Heights, California
  - Research Site, Inglewood, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, San Dimas, California
  - Research Site, West Covina, California
  - Research Site, Whittier, California
  - Research Site, Pembroke Pines, Florida
  - Research Site, Blairsville, Georgia
  - Research Site, East Point, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Quincy, Illinois
  - Research Site, Columbia, Mississippi
  - Research Site, Pachuta, Mississippi
  - Research Site, Lincoln, Nebraska
  - Research Site, Livingston, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Maspeth, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, King, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Yadkinville, North Carolina
  - Research Site, Arlington, Texas
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, South Charleston, West Virginia
- Research Site, San Juan, Puerto Rico

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 16 June 2010 through 02 July 2012, 2248 participants were enrolled in the study. A total of 51 small dialysis organization facilities enrolled in the study, of these, 45 (88.2%) facilities reported completing the study, 5 (9.8%) discontinued and 1 site was unaccounted for.
Period: Overall Study
Arm/Group | Cohort
Started | 2248
Completed | 1182
Not Completed | 1066
Not completed — Ineligibility determined | 6
Not completed — Protocol deviation | 6
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 11
Not completed — Death | 439
Not completed — Protocol-specified criteria | 551
Not completed — Other | 40

BASELINE CHARACTERISTICS:
Arm/Group | Cohort
Number analyzed (Participants) | 2248
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 966
  Male | 1282
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 7
  Asian/Pacific Islander | 258
  Black or African American | 557
  White | 1246
  Other | 171
  Unknown | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 646
  Neither Hispanic or Latino | 1602
Dialysis modality at enrollment [Number; unit: participants]
  Peritoneal | 125
  Hemodialysis (in center) | 2107
  Home hemodialysis | 13
  Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Per Facility With Hemoglobin < 10 g/dL
Description: The percentage of participants within each small dialysis organization (SDO) facility with hemoglobin < 10 g/dL over time. Percentage of participants meeting the criteria at the facility-level were calculated for each facility first and then summarized across facilities as a continuous variable, weighted by the number of participants in a facility.
Time Frame: Data were collected monthly from June 2010 until September 2012
Population: Facilities with at least one non-missing hemoglobin record for participants included in the primary analysis set (all enrolled participants) at each time point (indicated by n).
Measure: Mean (95% Confidence Interval); unit: percentage of participants per facility
Units Other Than Participants: SDO facilities
Arm/Group | Cohort
Number analyzed (Participants) | 2248
Number analyzed (SDO facilities) | 51
percentage of participants per facility
  June 2010 (n=39) | 11.5 [9.4 to 13.6]
  July 2010 (n=45) | 11.0 [8.3 to 13.8]
  August 2010 (n=50) | 13.1 [10.9 to 15.0]
  September 2010 (n=51) | 12.0 [10.0 to 13.9]
  October 2010 (n=51) | 12.7 [11.1 to 14.2]
  November 2010 (n=51) | 13.2 [11.3 to 15.0]
  December 2010 (n=51) | 14.3 [11.9 to 16.4]
  January 2011 (n=50) | 13.5 [11.6 to 15.3]
  February 2011 (n=50) | 18.3 [15.6 to 21.0]
  March 2011 (n=50) | 16.4 [13.7 to 19.3]
  April 2011 (n=50) | 16.9 [13.8 to 19.8]
  May 2011 (n=50) | 15.4 [12.7 to 18.2]
  June 2011 (n=50) | 16.7 [14.0 to 19.3]
  July 2011 (n=50) | 14.0 [11.9 to 16.1]
  August 2011 (n=50) | 15.5 [13.2 to 17.8]
  September 2011 (n=50) | 19.3 [16.6 to 22.4]
  October 2011 (n=50) | 21.7 [18.7 to 25.2]
  November 2011 (n=50) | 22.2 [18.8 to 25.6]
  December 2011 (n=48) | 21.8 [18.7 to 25.7]
  January 2012 (n=48) | 22.0 [18.2 to 26.4]
  February 2012 (n=48) | 19.5 [15.9 to 23.8]
  March 2012 (n=48) | 23.3 [19.7 to 27.1]
  April 2012 (n=48) | 24.0 [20.8 to 27.3]
  May 2012 (n=48) | 25.1 [21.1 to 28.9]
  June 2012 (n=45) | 24.6 [20.7 to 29.1]
  July 2012 (n=45) | 23.1 [20.2 to 26.8]
  August 2012 (n=45) | 22.6 [19.2 to 26.4]
  September 2012 (n=45) | 22.2 [17.8 to 26.6]

2. Secondary Outcome: Percentage of Participants Treated by Each Dialysis Modality
Description: The percentage of participants treated with peritoneal, hemodialysis (in center) or home hemodialysis over the course of the study. For participants who switched modalities within a quarter, the last current modality is reported.
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point
Measure: Number; unit: percentage of participants
Groups:
- Q4 2010: Fourth quarter (Q4) 2010
- Q1 2011: First quarter (Q1), 2011
- Q2 2011: Second quarter (Q2), 2011
- Q3 2011: Third quarter (Q3) 2011
- Q4 2011: Fourth quarter, 2011
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1819 | 1810 | 1701 | 1646 | 1554
percentage of participants
  Peritoneal | 2.0 | 2.2 | 3.6 | 2.8 | 2.9
  Hemodialysis (in center) | 94.4 | 93.0 | 93.0 | 92.6 | 93.0
  Home hemodialysis | 0.5 | 0.7 | 0.6 | 0.7 | 0.6
  Missing | 3.0 | 4.2 | 2.8 | 3.9 | 3.5

3. Primary Outcome: Percentage of Participants Per Facility With Hemoglobin > 12 g/dL
Description: The percentage of participants within each small dialysis organization (SDO) facility with hemoglobin > 12 g/dL over time. Percentage of participants meeting the criteria at the facility-level were calculated for each facility first and then summarized across facilities as a continuous variable, weighted by the number of participants in a facility.
Time Frame: Data were collected monthly from June 2010 until September 2012
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants per facility
Units Other Than Participants: SDO facilities
Arm/Group | Cohort
Number analyzed (Participants) | 2248
Number analyzed (SDO facilities) | 51
percentage of participants per facility
  June 2010 (n=39) | 30.2 [25.4 to 35.5]
  July 2010 (n=45) | 28.3 [25.1 to 31.6]
  August 2010 (n=50) | 28.2 [25.2 to 31.5]
  September 2010 (n=51) | 30.6 [27.7 to 34.0]
  October 2010 (n=51) | 28.7 [26.4 to 31.3]
  November 2010 (n=51) | 27.8 [24.9 to 30.8]
  December 2010 (n=51) | 24.5 [22.1 to 27.2]
  January 2011 (n=50) | 25.6 [22.7 to 29.0]
  February 2011 (n=50) | 24.5 [21.4 to 28.1]
  March 2011 (n=50) | 22.8 [19.6 to 26.2]
  April 2011 (n=50) | 21.8 [18.7 to 25.5]
  May 2011 (n=50) | 23.2 [20.2 to 26.7]
  June 2011 (n=50) | 18.5 [15.5 to 22.2]
  July 2011 (n=50) | 20.2 [17.3 to 23.6]
  August 2011 (n=50) | 19.0 [16.3 to 22.0]
  September 2011 (n=50) | 18.2 [15.6 to 21.2]
  October 2011 (n=50) | 14.3 [12.3 to 16.3]
  November 2011 (n=50) | 11.5 [9.8 to 13.3]
  December 2011 (n=48) | 11.8 [9.8 to 13.7]
  January 2012 (n=48) | 13.7 [11.8 to 15.9]
  February 2012 (n=48) | 12.5 [10.4 to 15.3]
  March 2012 (n=48) | 11.2 [9.4 to 13.1]
  April 2012 (n=48) | 10.3 [8.7 to 12.2]
  May 2012 (n=48) | 11.6 [9.6 to 13.7]
  June 2012 (n=45) | 12.1 [10.1 to 14.2]
  July 2012 (n=45) | 11.9 [9.4 to 14.5]
  August 2012 (n=45) | 11.6 [9.4 to 13.9]
  September 2012 (n=45) | 13.1 [10.9 to 15.3]

4. Primary Outcome: Percentage of Participants Per Facility With Urea Reduction Ratio (URR) ≥ 65%
Description: The percentage of participants within each small dialysis organization (SDO) facility with a urea reduction ratio ≥ 65% over time. URR is calculated as:
  Baseline urea level - post-baseline urea level/baseline urea level * 100. Percentage of participants meeting the criteria at the facility-level were calculated for each facility first and then summarized across facilities as a continuous variable, weighted by the number of participants in a facility.
Time Frame: Data were collected monthly from June 2010 until September 2012
Population: Facilities with at least one non-missing URR record for participants included in the primary analysis set (all enrolled participants) at each time point (indicated by n).
Measure: Mean (95% Confidence Interval); unit: percentage of participants per facility
Units Other Than Participants: SDO facilities
Arm/Group | Cohort
Number analyzed (Participants) | 2248
Number analyzed (SDO facilities) | 51
percentage of participants per facility
  June 2010 (n=37) | 84.8 [81.4 to 88.3]
  July 2010 (n=44) | 85.0 [81.5 to 88.5]
  August 2010 (n=49) | 85.0 [82.5 to 87.5]
  September 2010 (n=50) | 86.9 [84.3 to 89.5]
  October 2010 (n=50) | 87.9 [85.2 to 90.3]
  November 2010 (n=50) | 87.8 [85.2 to 90.3]
  December 2010 (n=50) | 86.9 [84.3 to 89.3]
  January 2011 (n=49) | 85.5 [82.1 to 88.7]
  February 2011 (n=49) | 86.7 [83.9 to 89.4]
  March 2011 (n=49) | 88.4 [86.1 to 90.6]
  April 2011 (n=49) | 87.8 [85.5 to 90.0]
  May 2011 (n=49) | 88.8 [85.9 to 91.4]
  June 2011 (n=49) | 90.2 [88.3 to 92.0]
  July 2011 (n=49) | 89.0 [87.0 to 90.9]
  August 2011 (n=49) | 89.0 [86.9 to 91.0]
  September 2011 (n=49) | 89.5 [87.6 to 91.6]
  October 2011 (n=49) | 90.4 [88.1 to 92.4]
  November 2011 (n=49) | 89.2 [86.0 to 91.9]
  December 2011 (n=47) | 90.3 [88.0 to 92.4]
  January 2012 (n=47) | 88.7 [86.1 to 91.2]
  February 2012 (n=47) | 89.3 [86.9 to 91.5]
  March 2012 (n=48) | 89.4 [87.0 to 91.7]
  April 2012 (n=47) | 90.9 [88.4 to 93.5]
  May 2012 (n=47) | 91.1 [89.1 to 93.1]
  June 2012 (n=44) | 91.1 [89.0 to 92.9]
  July 2012 (n=44) | 91.3 [88.9 to 93.4]
  August 2012 (n=44) | 91.4 [88.8 to 94.0]
  September 2012 (n=44) | 93.3 [91.6 to 95.0]

5. Secondary Outcome: Percentage of Participants in Each Vascular Access Type Category
Description: The percentage of participants in each vascular access type category out of all enrolled participants on hemodialysis over the course of the study.
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study and on hemodialysis at each time point
Measure: Number; unit: percentage of participants
Groups:
- Q4 2010: Fourth quarter, 2010
- Q1 2011: First quarter 2011
- Q2 2011: Second quarter, 2011
- Q3 2011: Third quarter, 2011
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1718 | 1683 | 1582 | 1524 | 1445
percentage of participants
  Arteriovenous fistula | 62.8 | 63.2 | 63.5 | 63.8 | 63.7
  Arteriovenous graft | 17.2 | 16.8 | 16.2 | 16.0 | 15.5
  Venous catheter | 19.9 | 20.0 | 20.2 | 20.1 | 20.7
  Missing | 0.1 | 0.1 | 0.1 | 0.1 | 0.1

6. Secondary Outcome: Percentage of Participants Per Facility Receiving Erythropoietin Stimulation Agents (ESA)
Description: The percentage of participants who received erythropoietin stimulation agents (ESA) in a facility over the course of the study. Mean and confidence interval (CI) are calculated across facilities and by using total number of participants actively receiving chronic dialysis in each facility per month as weight.
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set facilities / participants on study at each time point.
Measure: Mean (95% Confidence Interval); unit: percentage of participants per facility
Units Other Than Participants: Facilities
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1819 | 1810 | 1701 | 1646 | 1554
Number analyzed (Facilities) | 50 | 48 | 49 | 49 | 47
percentage of participants per facility | 91.2 [87.0 to 94.5] | 92.0 [89.1 to 94.5] | 90.9 [87.7 to 93.7] | 91.2 [88.5 to 94.0] | 89.4 [86.4 to 92.2]

7. Secondary Outcome: Percentage of Participants Receiving Cinacalcet
Description: The percentage of participants receiving cinacalcet (Sensipar) over time
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1819 | 1810 | 1701 | 1646 | 1554
percentage of participants | 22.3 | 26.2 | 29.3 | 30.0 | 31.0

8. Secondary Outcome: Percentage of Participants Receiving Phosphate Binding Agents
Description: The percentage of participants receiving phosphate binding agents over time
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1819 | 1810 | 1701 | 1646 | 1554
percentage of participants | 60.9 | 66.0 | 70.4 | 74.2 | 73.3

9. Secondary Outcome: Percentage of Participants Receiving a Vitamin D Sterol
Description: The percentage of participants receiving a vitamin D sterol (ie, calcitriol, alfacalcidol, paricalcitol or doxercalciferol) over time. Note that participants could receive more than one type of vitamin D sterol.
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1819 | 1810 | 1701 | 1646 | 1554
percentage of participants
  Any Vitamin D sterol | 80.6 | 76.2 | 77.5 | 77.7 | 79.4
  Intravenous | 76.0 | 68.0 | 66.5 | 62.6 | 62.7
  Oral - activated | 7.6 | 10.3 | 15.3 | 16.2 | 17.7
  Oral - not activated | 2.3 | 5.9 | 6.7 | 9.1 | 9.7

10. Secondary Outcome: Mean Hemoglobin Concentration by Quarter
Time Frame: Fourth quarter (Q4) 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point and with available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Q4 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1797 | 1773 | 1675 | 1610 | 1525
g/dL | 11.28 (1.35) | 11.17 (1.35) | 11.06 (1.25) | 11.00 (1.32) | 10.78 (1.22)

11. Secondary Outcome: Distribution of Facilities With Percentage of Participants With Hemoglobin < 10 g/dL Over Time
Description: Facilities were categorized over time based on the percentage of participants at the facility with hemoglobin < 10 g/dL: Faciities with 0 to <5% of participants with hemoglobin < 10 g/dL; Facilities with 5 to < 10% of participants with hemoglobin < 10 g/dL; Facilities with 10 to < 15% participants with hemoglobin < 10 g/dL; Facilities with 15 to < 20% of participants with hemoglobin < 10 g/dL; Facilities with ≥ 20% of participants with hemoglobin < 10 g/dL.
Time Frame: December 2010, March 2011, June 2011, September 2011, December 2011
Population: Facilities with at least one non-missing hemoglobin record, for participants included in the primary analysis set who were on study and with available data at each time point.
Measure: Number; unit: percentage of facilities
Units Other Than Participants: Facilities
Arm/Group | December 2010 | March 2011 | June 2011 | September 2011 | December 2011
Number analyzed (Participants) | 1789 | 1661 | 1592 | 1511 | 1420
Number analyzed (Facilities) | 51 | 50 | 50 | 50 | 48
percentage of facilities
  0%-<5% of participants with hemoglobin < 10 g/dL | 11.8 (1.36) | 10.0 (1.33) | 10.0 (1.23) | 4.0 (1.29) | 6.3 (1.21)
  5%-<10% of participants with hemoglobin <10 g/dL | 21.6 | 22.0 | 20.0 | 16.0 | 8.3
  10%-<15% of participants with hemoglobin <10 g/dL | 29.4 | 24.0 | 20.0 | 18.0 | 16.7
  15%-<20% of participants with hemoglobin <10 g/dL | 11.8 | 18.0 | 10.0 | 20.0 | 16.7
  ≥20% of participants with hemoglobin <10 g/dL | 25.5 | 26.0 | 40.0 | 42.0 | 52.1

12. Secondary Outcome: Percentage of Participants Per Facility With Transferrin Saturation < 20% and Ferritin Level < 100 ng/mL
Description: The mean percentage of participants per facility with transferrin saturation < 20% and ferritin level < 100 ng/mL. Mean and CI are calculated across facilities and by using number of participants with non-missing transferrin saturation and ferritin in each facility as weight.
Time Frame: December 2010, March 2011, June 2011, September 2011, December 2011
Population: Facilities / participants with at least one non-missing transferrin saturation or ferritin record at each time point.
Measure: Mean (95% Confidence Interval); unit: percentage of participants per facility
Units Other Than Participants: Facilities
Arm/Group | December 2010 | March 2011 | June 2011 | September 2011 | December 2011
Number analyzed (Participants) | 1399 | 1132 | 1160 | 1128 | 1064
Number analyzed (Facilities) | 46 | 43 | 44 | 43 | 40
percentage of participants per facility | 2.4 (1.36) [1.5 to 3.5] | 0.6 (1.33) [0.2 to 1.1] | 1.4 (1.23) [0.2 to 3.0] | 1.0 (1.29) [0.4 to 1.7] | 0.7 (1.21) [0.3 to 1.2]

13. Secondary Outcome: Cumulative Monthly Dose of Epoetin Alfa Administered
Description: The cumulative monthly intravenous epoetin alfa dose in participants on hemodialysis.
Time Frame: December 2010, March 2011, June 2011, September 2011, December 2011
Population: Primary Analysis Set participants on study and on hemodialysis and receiving epoetin alfa at each time point and with available data.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | December 2010 | March 2011 | June 2011 | September 2011 | December 2011
Number analyzed (Participants) | 1172 | 1188 | 1105 | 1096 | 984
units | 39000.0 [19100.0 to 71500.0] | 35000.0 [16650.0 to 66000.0] | 33800.0 [15400.0 to 65000.0] | 28000.0 [13000.0 to 52000.0] | 32900.0 [16000.0 to 60000.0]

14. Secondary Outcome: Number of Participants Taking Epoetin Alfa by Month
Description: The number of participants who took epoetin alfa only, by month, in participants on hemodialysis.
Time Frame: December 2010, March 2011, June 2011, September 2011, December 2011
Population: Primary Analysis Set participants on study and on hemodialysis at each time point.
Measure: Number; unit: participants
Arm/Group | December 2010 | March 2011 | June 2011 | September 2011 | December 2011
Number analyzed (Participants) | 1645 | 1566 | 1499 | 1421 | 1342
participants | 1269 (57684.5) | 1299 (52423.4) | 1244 (51344.7) | 1212 (48175.3) | 1140 (47792.1)

15. Secondary Outcome: Number of Participants With Transfusions, Hospitalizations, Mortality, and Transfers Out
Time Frame: June to December 2010, Q1 2011, Q2 2011, Q3 2011, and Q4 2011.
Population: Primary Analysis Set participants on study at each time point
Measure: Number; unit: participants
Groups:
- 2010: From June through December 2010
Arm/Group | 2010 | Q1 2011 | Q2 2011 | Q3 2011 | Q4 2011
Number analyzed (Participants) | 1873 | 1810 | 1701 | 1646 | 1554
participants
  Participants with transfusions | 54 | 56 | 50 | 39 | 36
  Participants who died | 71 | 67 | 52 | 55 | 46
  Participants with hospitalizations | 574 | 445 | 354 | 296 | 275
  Participants who transferred out | 63 | 51 | 31 | 47 | 21

ADVERSE EVENTS:
Time Frame: Up to 28 months
Description: As this was a non-interventional observational study, only serious adverse drug reactions (SADRs) relating to Amgen products were reported. An adverse drug reaction (ADR) was defined for this study as any undesirable experience or worsening of a pre-existing medical condition associated with the use of a medicine in a clinical study participant.
Arm/Group | Cohort
Serious Adverse Events (participants affected / at risk) | 1/2248
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort (N=2248)
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.